CLINICAL TRIAL: NCT02277197
Title: A Phase 1b Study of Ficlatuzumab and Cetuximab in Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma With Biomarker Correlatives
Brief Title: Ficlatuzumab and Cetuximab in Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: James J Lee (Other)
Collaborators: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, James J Lee, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13-059
Record Dates: First submitted 2014-10-25; First posted 2014-10-28 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck; Squamous Cell Carcinoma of the Head and Neck; Squamous Cell Carcinoma, Head And Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — ficlatuzumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ficlatuzumab and Cetuximab (Experimental): Ficlatuzumab will be administered as an IV infusion over 30-60 minutes, once every 2 weeks. Ficlatuzumab will be administered 30-60 minutes after the completion of the cetuximab infusion.
  Cetuximab will be administered as an IV infusion once every 2 weeks. The first dose will be administered over 120 minutes (± 15 minutes). Subsequent doses may be infused over 60 minutes (± 15 minutes). The starting dose of cetuximab (dose tier 1) will be 500 mg/m2. Cetuximab will be administered prior to ficlatuzumab.
  Interventions: Drug: Ficlatuzumab; Drug: Cetuximab

INTERVENTIONS:
Drug: Ficlatuzumab — Ficlatuzumab Concentrate for Injection, 20 mg/mL, is formulated in 10 mM histidine buffer pH 5.8. The formulation also includes 142 mM arginine (for isotonicity) and 0.01% polysorbate 80. The product is sterile filtered and aseptically filled into washed and depyrogenated 5 mL glass vials.The product is a clear to slightly opalescent, colorless to slightly yellow, solution.
  Ficlatuzumab Concentrate for Injection is to be administered by IV infusion as an admixture with normal saline solution. The admixture solution in an IV bag is connected to an infusion set containing a 0.22 µm low protein-binding in line filter. The filtered admixture solution is clear to slightly opalescent.
  Ficlatuzumab is to be stored under refrigerated conditions (2o C- 8oC)
  Other Names: AV-299; SCH 900 105
Drug: Cetuximab — Cetuximab is supplied as a 50-mL, single-use vial containing 100 mg of cetuximab at a concentration of 2 mg/mL in phosphate buffered saline. The solution should be clear and colorless and may contain a small amount of easily visible white amorphous cetuximab particulates. Cetuximab can be administered via infusion pump or syringe pump, it must not be administered as an IV push or bolus. Cetuximab must be administered with the use of a low protein binding 0.22-micrometer in-line filter. Maximum infusion rate should not exceed 5 mL/min.
  Store vials under refrigeration at 2C to 8C (36F to 46F). DO NOT FREEZE. Following the cetuximab infusion, a one-hour observation period is recommended.
  Other Names: Erbitux; IMC-C225; C225; CAS number: 205923-56-4; Lilly compound number: LY2939777; Chemical name: Chimeric anti-EGFR antibody

SUMMARY:
The epidermal growth factor receptor (EGFR) is both oncogene and prognostic biomarker in head and neck squamous cell carcinoma (HNSCC). EGFR's functional importance in HNSCC resulted in development of the first molecularly targeted strategy, the anti-EGFR monoclonal antibody cetuximab. Given the lack of therapeutic options for patients with recurrent/metastatic HNSCC after failure of cetuximab, there is strong scientific interest in understanding resistance in order to identify new therapies for this population. A possible resistance mechanism to anti-EGFR therapy in HNSCC is primary or compensatory activation of alternate growth factor receptors including c-Met. The MET oncogene encodes c-Met, an RTK bound exclusively by the ligand, hepatocyte growth factor (HGF). The HGF/c-Met signaling pathway converges with the EGFR network at both the PI3K/Akt and MAPK nodes. Laboratory data suggest the ability for reciprocal compensation between EGFR and c-Met. We hypothesize that HGF/c-Met pathway inhibition may overcome resistance to cetuximab in patients with HNSCC, such as those with clinical cetuximab resistance.

Ficlatuzumab (AV-299) is a humanized HGF-inhibitory immunoglobulin G1 (IgG1) monoclonal antibody. The primary objective of this phase 1b study is to find the recommended phase II dose (RP2D) of the combination of ficlatuzumab and cetuximab in patients with recurrent/metastaticHNSCC. The dose-finding study design will follow a Narayana k-in-a-row design with k set to 2 to target a 33% rate of dose-limiting toxicity (DLT). In the dose-finding phase, a total of 8 patients will be treated if no DLTs are observed or 14 patients if at least one DLT occurs. An expansion cohort will then proceed at RP2D until 12 patients have been treated at that dose level with the combination of ficlatuzumab and cetuximab. We will evaluate biomarkers of HGF/cMet pathway activation in baseline tissue, plasma and immune cells for a preliminary relationship with clinical activity.

DETAILED DESCRIPTION:
This is a phase 1b, single arm, open-labeled study of ficlatuzumab and cetuximab in recurrent/metastatic HNSCC with biomarker correlatives. The primary objective of this study is to establish the recommended-for-phase II dose (RP2D) of the combination of ficlatuzumab and Cetuximab. In the absence of treatment delays due to adverse event(s), treatment may continue until disease progression or until one of the following criteria applies:

* Disease progression,
* Intercurrent illness that prevents further administration of treatment,
* Unacceptable adverse event(s),
* Patient decides to withdraw from the study, or
* General or specific changes in the patients condition render the patient unacceptable for further treatment in the judgment of the investigator.

After progressive disease, subjects will be followed for survival every 3 months for 2 years.

Cetuximab and ficlatuzumab are administered every other week on day 1 and 15 of a 28-day cycle. Ficlatuzumab will be administered as an IV infusion, over 30-60 minutes,10 mg/kg every 2 weeks, on the same day as the first dose of cetuximab. Ficlatuzumab will be administered 30-60 minutes after the completion of the cetuximab infusion. Cetuximab will be administered prior to ficlatuzumab as an IV infusion. The first dose will be administered over 120 minutes (± 15 minutes). Subsequent doses may be infused over 60 minutes (± 15 minutes).The starting dose of cetuximab (dose tier 1) will be 500 mg/m2 every 2 weeks.

Subjects will be monitored for adverse events and toxicity during study treatment and for 30 days after last dose of ficlatuzumab. Blood will be drawn for correlative studies at baseline, and at the end of every even cycle. Prior to initiation of protocol treatment, patients will undergo a mandatory research biopsy.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Patients must have histologically confirmed HNSCC, from any primary site. Nasopharyngeal carcinoma, WHO Type I (keratinizing), will be included. Squamous cell carcinoma of unknown primary, clearly related to the head and neck, will be included.
* Recurrent/metastatic disease, fulfilling at least one of the criteria defined below:

  * Incurable disease as assessed by surgical or radiation oncology
  * Metastatic (M1) disease
  * Persistent or progressive disease following curative-intent radiation, and not a candidate for surgical salvage due to incurability or morbidity. Patients who decline radical surgery are eligible.
* In the dose-finding phase, patients may be cetuximab-exposed or cetuximab-naïve. If the most recent line of therapy included cetuximab, a two-week washout period without cetuximab dosing is required.
* Patients must have previously received, not tolerated, or been judged clinically unsuitable for platinum-containing therapy.
* In the dose-expansion phase, patients must be cetuximab-resistant by fulfilling at least one of the criteria defined below:

  * Disease recurrence within 6 months of completing definitive radiotherapy for locally advanced disease. Radiation must have included concurrent cetuximab. Induction chemotherapy, if given, may or may not have included cetuximab.
  * Disease progression during, or within 6 months, of cetuximab treatment in the recurrent/metastatic setting. Prior cetuximab exposure may have occurred in first, second and/or third line.
  * If the most recent line of therapy included cetuximab, a two-week washout period without cetuximab dosing is required.
* Eastern Cooperative Oncology Group Performance Status 0-1 at time of informed consent (see Appendix B)
* Age ≥ 18 years
* Patients must consent to a research biopsy of tumor tissue at baseline, for conduct of correlative studies. Archived biopsy material may not be substituted.
* Measurable disease per RECIST criteria, version 1.1 (see section 6)
* Patients must have the following laboratory values measured within 28 days of registration:

  * Absolute neutrophil count (ANC) ≥ 1500/mm3
  * Platelet count (PLT) ≥ 100,000/mm3
  * Creatinine clearance ≥ 40 ml/min as determined by 24-hour collection or estimated by the Cockraft-Gault formula:Calculated Creatinine Clearance = [(140-age) X (actual body weight in kg) X (0.85 if female)]/(72 X serum creatinine)
  * Serum bilirubin ≤ 1.5 times upper-limit of normal (ULN)
  * AST (aspartate aminotransferase) and ALT (alanine aminotransferase) ≤ 3 times ULN
* No prior severe infusion reaction to cetuximab or a monoclonal antibody
* Written informed consent must be obtained from all patients prior to beginning therapy. Patients should have the ability to understand and the willingness to sign a written informed consent document.
* If a woman of childbearing potential, documentation of negative pregnancy within 14 days prior to first dose of ficlatuzumab. Sexually active women of childbearing potential must agree to use adequate contraceptive measures, while on study and for 30 days after the last dose of study drug. All fertile female subjects (and their partners) must agree to use a highly effective method of contraception. Effective birth control includes (a) intrauterine device (IUD) plus one barrier method; or (b) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm).

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Nasopharyngeal primary site, if WHO Type II or III (non-keratinizing)
* History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational agent.
* Prior treatment with an HGF/cMet inhibitor such as rilotumumab, crizotinib, MetMAb, or ARQ197
* Uncontrolled central nervous system (CNS) metastases, including leptomeningeal metastases, are not allowed. Subjects with previously treated brain metastases will be allowed if the brain metastases have been stable without steroid treatment for at least 4 weeks following prior treatment (radiotherapy or surgery).
* Failure to recover to Grade 1 or baseline from all toxic effects of previous chemotherapy, radiation therapy, biologic therapy, and/or experimental therapy, with the exception of: alopecia, Grade ≤ 2 peripheral neuropathy, Grade ≤ 2 cetuximab-related rash or other skin changes, hypomagnesemia (acceptable values detailed below), hypokalemia (acceptable values detailed below), and the acceptable hematologic values summarized above. A washout period of 2 weeks from prior cetuximab is required; a washout period of 3 weeks from any prior cytotoxic chemotherapy or investigational drug is required.
* Significant pulmonary disease, including pulmonary hypertension or interstitial pneumonitis.
* Decreased serum albumin < 30 g/L (< 3 g/dL)
* Peripheral edema ≥ Grade 2 per NCI-CTCAE version 4.0.
* Significant electrolyte imbalance prior to enrollment (note that patients may be supplemented to achieve acceptable electrolyte values):

  * Hypomagnesemia <1.2 mg/dL or 0.5 mmol/L.
  * Hypocalcemia < 8.0 mg/dL or 2.0 mmol/L.
  * Hypokalemia < 3.0 mmol/L.
* Significant dermatological disease including, but not limited to, skin drying and fissuring, paronychial inflammation, infectious sequelae (eg, blepharitis, cheilitis, cellulitis, cyst). Exception: patients with Grade ≤ 2 cetuximab-related rash, xerosis, fissures or paronychial inflammation are eligible.
* Significant cardiovascular disease, including:

  * Cardiac failure New York Heart Association (NYHA) class III or IV.
  * Myocardial infarction, severe or unstable angina within 6 months prior to Study Day 1.
  * History of serious arrhythmia (i.e., ventricular tachycardia, or ventricular fibrillation).
  * Cardiac arrhythmias requiring anti-arrhythmic medications.
* Significant thrombotic or embolic events within 4 weeks prior to Study Day 1. Significant thrombotic or embolic events include but are not limited to stroke or transient ischemic attack (TIA). Catheter-related thrombosis is not a cause for exclusion. Diagnosis of deep vein thrombosis or pulmonary embolism is allowed if it occurred > 4 weeks prior to Study Day 1 and the patient is asymptomatic and stable on anti-coagulation therapy.
* Any other medical condition (eg, alcohol abuse) or psychiatric condition that, in the opinion of the Investigator, might interfere with the subject's participation in the trial or interfere with the interpretation of trial results.
* History of second malignancy within 2 years prior to Study Day 1 (except for excised and cured non-melanoma skin cancer, carcinoma in situ of breast or cervix, superficial bladder cancer, resected Stage I differentiated thyroid cancer, or T1a or T1b prostate cancer comprising < 5% of resected tissue with normal prostate specific antigen (PSA) since resection).
* Major surgery within 6 weeks prior to Study Day 1 (subjects must have completely recovered from any previous surgery prior to Study Day 1).
* Active infection requiring antibiotics or antifungals within 7 days prior to first dose of study drug.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible drug interactions with study drugs. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated. Note: HIV testing is not required for entry into this protocol.
* Women must not be pregnant or breastfeeding because ficlatuzumab and/or cetuximab may be harmful to the fetus or the nursing infant. Pregnant women are excluded from this study because ficlatuzumab and/or cetuximab have the potential for teratogenic or abortifacient effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Establish the recommended-for-phase II dose (RP2D) of the combination of ficlatuzumab and cetuximab. | 1 year
  A dose escalation/de-escalation plan will be conducted according to an adaptive Narayana k-in-a-row design.45 We will select the dose of ficlatuzumab that is close to but does not exceed a 33% dose limiting toxicity (DLT) rate when administered with a fixed q2week dose of cetuximab. The observation period for identifying a DLT will be the first cycle, which consists of two doses of ficlatuzumab, or 4 weeks.In the dose-finding phase, a total of 8 patients will be treated if no DLTs are observed or 14 patients if at least one DLT occurs. If no DLTs are observed among the first 8 patients, the recommended for phase 2 dose (RP2D) will be set to dose tier 2. If a DLT is observed and 14 patients are treated and observed, the RP2D will be estimated from DLTs across all dose levels by isotonic regression. More than one patient can be enrolled at the same time.

SECONDARY OUTCOMES:
Preliminary clinical efficacy of the combination of cetuximab and ficlatuzumab in patients with R/M HNSCC, including PFS, RR, and OS. | 5 year
  Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used.
  Progression-free survival (PFS) will be calculated from treatment initiation to disease progression or death from any cause or last follow up.
  Survival will be measured from the date of entry on study. The preliminary clinical efficacy of the combination of cetuximab and ficlatuzumab will be described according to RR, median PFS, and median OS in: 1) the entire study population; 2) patients with prior cetuximab exposure treated at RP2D.
Evaluate the relationship between tumor HGF and c-Met expression in baseline research biopsies and preliminary efficacy data | 5 years
  HNSCC tumors overexpress both HGF and c-Met as compared to adjacent tissue. The relationship of percent change in baseline sum diameter of index lesions to baseline cMet and HGF will be characterized by a linear, or if necessary, generalized linear or nonlinear regression model with appropriate confidence intervals.This exploratory endpoint seeks an early indication that overexpression of cMet or its ligand, HGF, may predict benefit from ficlatuzumab. For purposes of this endpoint, both cMet and HGF expression levels will be reported as semi-quantitative H-scores.
Describe biomarkers of HGF/c-Met and EGFR pathway activation in archived and baseline tumor biopsies | 5 years
  The prevalence of several mutations in HNSCC which interact with the HGF/c-Met signaling pathway have been identified, and may modulate the impact of pathway antagonism.These include PIK3CA (8%), PTEN (8%), and HRAS (4%) mutations.This will be evaluated by by whole exome sequencing.
Evaluate peripheral (blood) pharmacodynamic biomarkers of HGF/c-Met and EGFR pathway activation to correlate with preliminary efficacy data | 5 years
  Additional biomarkers in tumor and blood will be quantitatively measured and will be evaluated as predictors of tumor response and/or PFS in appropriate generalized linear models. Calculated p values for testing the significance of the prediction models will be adjusted for false discovery by the method of Benjamini and Hochberg
Describe dendritic and T cell phenotypes in archived and baseline tumor biopsies | 5 years
  HNSCC is an immunosuppressive disease. Patients demonstrate lower absolute lymphocyte counts than healthy subjects, impaired natural killer (NK) cell activity and poor antigen-presenting function. Mechanistically, HGF inhibits dendritic cell activation. Dendritic cell and T cell phenotypes will be evaluated in archived biopsies (prior to cetuximab resistance) and pre ficlatuzumab research biopsies.
Evaluate pharmacodynamic biomarkers of peripheral T cell and NK cell activation to correlate with preliminary efficacy data | 5 years
  Additional biomarkers in tumor and blood will be quantitatively measured and will be evaluated as predictors of tumor response and/or PFS in appropriate generalized linear models. Calculated p values for testing the significance of the prediction models will be adjusted for false discovery by the method of Benjamini and Hochberg.Peripheral T cell and NK cell activity will be analyzed longitudinally before, during and after exposure to ficlatuzumab.
Describe toxicity and patient-reported quality of life | 5 years
  All patients will be evaluable for toxicity from the time of their first treatment with ficlatuzumab. The proportion of DLTs in each dosing cohort will be reported, as will the proportion of AEs in accordance with NCI CTCAE v.4 grading criteria.

CONTACTS AND LOCATIONS:
Overall Officials: James Ohr, DO, Principal Investigator — Attending Physician, UPMC Hillman Cancer Center
Locations (3):
- United States (3):
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Shadyside, Pittsburgh, Pennsylvania